CLINICAL TRIAL: NCT01269983
Title: Effectiveness of Fascial Manipulation for Chronic Low Back Pain. A Randomized Controlled Trial
Brief Title: Effectiveness of Fascial Manipulation for Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Mirco Branchini - Dr. Physioterapist, Degree Course in Physiotherapy - University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CdL_Ft_lombalgia_09
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2009-04

CONDITIONS: Low Back Pain
Keywords: low back pain; fascial manipulation; physioterapy; physical activity
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fascial manipolation (Experimental): 8 treatment sessions: 4 of fascial manipulation treatment, and 4 of standard physiotherapy (rexing exercise, stretching, abdominal and paravertebral isometric muscular recruiting)
  Interventions: Other: Fascial Manipulation
- physiotherapy (Active Comparator): 8 treatment sessions of standard physiotherapy (rexing exercise, stretching, abdominal and paravertebral isometric muscular recruiting)
  Interventions: Other: Fascial Manipulation

INTERVENTIONS:
Other: Fascial Manipulation — 8 treatment session in 4 weeks: every week both fascial manipulation and standard physiotherapy
  Other Names: manipolazione fasciale; manipolazione della fascia; manipulacion de la fascia

SUMMARY:
The purpose is to evaluate the effectiveness of a physiotherapy program for chronic low back pain. We'll randomize more about 35 patients in two groups. Both groups will receive an 8 physioterapy intervention in 4 weeks, in particular the first group (study) will receive 4 Fascial Manipulation treatment combined with 4 session of a standard approach (mobilization and stretching exercises); whereas the second (control) will receive only the standard approach.

DETAILED DESCRIPTION:
All patients were assessed and randomised by a physician. The control group intervention concerned of: relaxation of lumbar and respiration muscles, stretching for posterior muscular chain and hip flexors, assisted/active mobilization of lumbar region in sagittal plane and rotation, exercises to improve proprioception of lumbar spine, active and progressive movement of lumbar spine in anterior flexion, extension, lateroflexion and rotation, active exercise for lumbar stabilizers muscles, occupational training for activity of daily living, indications and recommendations for correct postures. The study group intervention received 4 manual intervention on deep fascial tissues, according to fascial manipulation tecnique, providing a specific motor and manual assessment, and a deep manual intervention over specific fascial alteration.

ELIGIBILITY:
Inclusion Criteria:

* patients with a chronic low back pain (more than 7 weeks)
* age between 20 to 60 years old

Exclusion Criteria:

* presence of neurological red flags
* continuative assumption of drugs for low back pain
* no positive imaging for spine lesions (fractures, spondilolistesi,
* vascular desease (aneurism abdominal aorta)
* secondary lesions (oncological desease)
* rheumatic systemic desease
* any other neurological desease which could compromise the partecipation to the program exercise

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
disabilty level, evaluated with the Roland and Morris Disability Questionnaire | from the first evaluation, at the end of the treatment
  we'll compare the baseline data (the first evaluation), with data at the end of the treatment, and with at every fullow up (30 and 90 days from the end of the treatment)

SECONDARY OUTCOMES:
pain and social activity level evaluated with Brief Pain Inventory. | from the first evaluation, at the end of the treatment
  we'll compare the baseline data (the first evaluation), with data at the end of the treatment, and with at every fullow up (30 and 90 days from the end of the treatment)
quality of life, evaluated with SF-36 | from the first evaluation, at the end of the treatment
  we'll compare the baseline data (the first evaluation), with data at the end of the treatment, and with at every fullow up (30 and 90 days from the end of the treatment)
pain, assessed with visual analogical scale | at the first evaluation, at the end of the treatment
  we'll compare the baseline data (the first evaluation), with data at the end of the treatment, and with at every fullow up (30 and 90 days from the end of the treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Mirco Branchini, Ph., Study Director — University of Bologna - Degree course in Physioterapy
Locations (1):
- Universitary Hospital of Bologna - S.Orsola Malpighi, Bologna, Italy

REFERENCES:
- [Background] Langevin HM, Stevens-Tuttle D, Fox JR, Badger GJ, Bouffard NA, Krag MH, Wu J, Henry SM. Ultrasound evidence of altered lumbar connective tissue structure in human subjects with chronic low back pain. BMC Musculoskelet Disord. 2009 Dec 3;10:151. doi: 10.1186/1471-2474-10-151. PMID 19958536
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Bednar DA, Orr FW, Simon GT. Observations on the pathomorphology of the thoracolumbar fascia in chronic mechanical back pain. A microscopic study. Spine (Phila Pa 1976). 1995 May 15;20(10):1161-4. doi: 10.1097/00007632-199505150-00010. PMID 7638659
- See also: This is the official link of Fascial Manipulation tecnique — http://fascialmanipulation.com